CLINICAL TRIAL: NCT06968312
Title: Testing Potential Enhancement of Standard Cognitive Processing Therapy for PTSD Using Hexadecanal: A Randomized Controlled Trial
Brief Title: Hexadecanal as an Addon to Cognitive Processing Therapy for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor of Psychology and Neuroscience, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HEX-PTSD
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Post Traumatic Stress Disorder (PTSD)
Keywords: PTSD; Posttraumatic Stress Disorder; Hexadecanal; treatment; CPT; Cognitive Processing Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — hexadecanal

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assign in a 1:1 ratio to either the active (HEX) or mineral oil (control) conditions.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The randomization list is prepared in advance. Research assistants with no contact with the patients, therapists, or independent clinical assessors operate the odor dispensers according to the randomization schedule in the designated rooms where treatments take place.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEX (Active Comparator): Participants with PTSD who undergo Cognitive Processing Therapy will receive Hexadecanal molecules diffused in the therapy room.
  Interventions: Other: Cognitive Processing Therapy + Hexadecanal; Other: Hexadecanal - Molecule Distribution in the Therapy room
- Control (Placebo Comparator): Participants with PTSD who undergo Cognitive Processing Therapy will receive control mineral oil molecules diffused in the therapy room.
  Interventions: Other: Cognitive Processing Therapy + Hexadecanal; Other: Hexadecanal - Molecule Distribution in the Therapy room

INTERVENTIONS:
Other: Cognitive Processing Therapy + Hexadecanal — Cognitive Processing Therapy is a protocolized, trauma-focused, CBT type treatment for PTSD.
Other: Hexadecanal - Molecule Distribution in the Therapy room — Distribution of a naturally secreted molecule from body odor (Hexadecanal).

SUMMARY:
This RCT investigates whether Cognitive Processing Therapy, a first line treatment for PTSD, can be enhanced by the use of the odor molecule Hexadecenal (HEX). HEX is secreted from body odor and has been shown to promotes psychological well-being and positive social interaction. For the active group Hex will be diffused in the treatment room during all treatment sessions. For the control group a vehicle placebo molecule will be diffused. Both therapists and patients will be blind to study condition.

DETAILED DESCRIPTION:
In this triple blind (patient, therapist, independent evaluator) RCT, 40 patients with PTSD receiving standard Cognitive Processing Therapy will be randomized in a 1:1 ratio to receive either odorless Hexadecanal molecules or odorless mineral oil molecules (Control) diffused in the treatment room at all therapy sessions. Inclusion criteria: age>18 years, PTSD diagnosis according to DSM-5-TR. Exclusion: Bipolar, psychotic, or neurological disorders, drug abuse, any parallel psychotherapy, anosmia. Primary outcome: pre-to-post treatment change in PTSD symptom severity measured by the PTSD check List for DSM-5 (PCL-5). Additional outcomes: Depression (PHQ-9), anxiety (GAD-7), Anger (DAR-5), therapeutic alliance (WAI-SF).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD according to DSM-5
* Age 18 years and over
* Eligible for CPT treatment at the National Center for Traumatic Stress and Resilience

Exclusion Criteria:

* Bipolar disorder, psychosis, neurological disorders
* Drug Addiction
* Parallel psychotherapy
* Congenital or acquired anosmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist (PCL-5) | 12-16 weeks
  A 20-item self-reported questionnaire on PTSD symptoms according to DSM-5

SECONDARY OUTCOMES:
Patient Health Questionnaire - 9 (PHQ-9) | 12-16 weeks
  A 9-item self-reported questionnaire on depression symptoms according to DSM-5
Generalized Anxiety Disorder -7 (GAD-7) | 12-16 weeks
  A 7-item self-reported questionnaire on generalized anxiety
Dimensions of Anger Reactions - 5 (DAR-5) | 12-16 weeks
  A 5-item self-reported questionnaire on anger
Working Alliance Inventory Short Form (WAI-SF | 12-16 weeks
  Completed by patent and therapist - ranks the quality of therapeutic alliance

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar Haim, PhD, Principal Investigator — Tel Aviv University; Noam Sobel, PhD, Study Director — Weizmann Institute of Science
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Endevelt-Shapira, Y. (2018). The role of chemosignaling in human social interaction (Doctoral dissertation, The Weizmann Institute of Science (Israel).